CLINICAL TRIAL: NCT05132348
Title: Immunological Markers for the Improvement of Diagnosis and Therapy of Osteoporosis
Brief Title: Immunophenotyping in Patients With Osteoporosis
Acronym: IPO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, PD Dr. Andreas Strauß, PD. Dr. med., University Hospital, Bonn
Other Study IDs: IPO15102021
Record Dates: First submitted 2021-10-20; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Immunophenotyping Blood Samples of Patients With Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples of patients with osteoporosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Immunological markers — Markers of blood samples of patients suffering from osteoporosis will be analyzed

SUMMARY:
In addition to a medical history and clinical examination, the diagnosis of osteoporosis includes the measurement of bone surface density by means of dual X-ray absorptiometry (DXA). In addition, blood tests are performed for certain parameters, such as vitamin D, calcium, phosphate and C-reactive protein. In order to optimize osteoporosis diagnostics, the development of further specific methods is required. The modulation of the immune system seems promising in this respect, since osteoporosis is based on an inflammatory reaction. Various regulatory markers of the innate and acquired immune system, which seem to be relevant in the development of the disease, have already been detected in osteoporosis patients. This study may help to gain new insights into disease-associated immunoregulatory markers that could revolutionize both the diagnosis and therapy of osteoporosis in the long term. By means of a simple blood test, patients could be diagnosed early and without additional radiation exposure, and effective therapy options could be developed.

DETAILED DESCRIPTION:
Osteoporosis is a disease of bone metabolism. The underlying disturbance of bone homeostasis promotes bone fractures and, in advanced stages, especially spontaneous fractures. The diagnosis of osteoporosis is carried out as part of routine clinical practice. In addition to the patient's medical history and clinical examination, blood tests are also carried out on certain parameters, including the concentrations of vitamin D, calcium and phosphate as well as C-reactive protein. In addition, bone density is measured by dual X-ray absorptiometry (DXA). The results can be used to determine the degree of osteoporosis, which affects the further therapeutic approach.

Therapy is essentially based on fracture prevention through optimization of dietary habits, promotion of physical activity, and adequate vitamin D intake. Pharmacological options mainly do not counteract the pathological bone loss and are usually not tolerable due to serious side effects or are only approved for a limited period of use. Consequently, the development of further options to complement existing methods is required for the diagnosis and treatment of osteoporosis. The modulation of the immune system seems to be promising, since osteoporosis is based on an inflammatory reaction. Thus, various regulatory markers of the innate and acquired immune system, which seem to be relevant in the development of the disease, have already been detected in osteoporosis patients. However, central questions regarding the immune phenotype of affected individuals remain unanswered. For example, it is unclear to what extent certain molecules, mostly growth factors or chemokines, influence the inflammatory processes in the context of osteoporosis. Furthermore, it is controversial whether and, if so, how immune markers influence each other and what effects this has on bone metabolism.In the long term, new insights regarding the properties of disease-associated immunoregulatory markers could revolutionize the diagnostic possibilities for osteoporosis, as affected individuals could be identified early and without additional radiation exposure by simple blood tests. Equally relevant is corresponding information for the improvement of therapy. In the future, the causative immune processes could be treated by regulating the corresponding immunological markers and meaningfully expand existing therapy options.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) diagnosed with osteoporosis.
* Written informed consent from the patient

Exclusion Criteria:

* Patients without diagnosed osteoporosis
* Patients without written informed consent
* Patients < 18 years old
* Patients with secondary osteoporosis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with diagnosed osteoporosis will be analyzed in this study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2026-02-19 (Estimated); Study Completion 2026-10-19 (Estimated)

PRIMARY OUTCOMES:
Immunological Marker | 2 hours
  Standardized values for the diagnosis of osteoporosis are examined in the blood samples taken. In addition, one serum sample and one EDTA sample (S-Monofat, Sarstedt AG & Co. KG, Nümbrecht, Germany, 7.5 ml each) are taken in order to analyze the immunophenotype on the cellular level as well as on the basis of soluble markers. Following the puncture, these samples are processed in the research laboratory of the Clinic for Orthopedics and Trauma Surgery and examined using various immunoassays.
DXA Values | 30 minutes
  Measurement of bone surface density using DXA scans

SECONDARY OUTCOMES:
Secondary Osteoporosis | 5 Minutes
  In addition to the medical history and clinical examination, all patients included in the study will complete a questionnaire to exclude a secondary form of osteoporosis. Among other things, previous occurrence of (spontaneous) fractures of the patients as well as the family history with regard to other diseases and fractures will be asked. The questionnaire is based on the S3 guideline of the German Osteoporosis Organization.
Menstruation | 2 Minutes
  Patients are also asked whether the measurements take place at the time of their menstruation.
Anthropometric Data | 3 Minutes
  Assessment of weight in kilograms, height in meters and age in years in form of questionnaire. Weight and height will be combined to report BMI in kg/m^2.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Strauß, PD Dr., Principal Investigator — physican
Locations (1):
- University Hospital of Bonn, Bonn, Northrhine Westfalia, Germany

IPD SHARING:
Plan to Share IPD: No